CLINICAL TRIAL: NCT00089869
Title: A Combination of Two Currently Approved Drugs to Enhance the Treatment of Schizophrenia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Purpose: Treatment
Other Study IDs: 8269; H6U-MC-HGLM
Record Dates: First submitted 2004-08-16; First posted 2004-08-18 (Estimated); Last update posted 2006-07-20 (Estimated); Status verified 2006-07

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Olanzapine; Atomoxetine Hydrochloride

INTERVENTIONS:
Drug: olanzapine
Drug: atomoxetine
Drug: placebo

SUMMARY:
Study of a medication for the treatment of Schizophrenia in patients who are already taking Abilify, Risperdal, Seroquel, Zyprexa

ELIGIBILITY:
Inclusion Criteria:

* Must have a clinical diagnosis of Schizophrenia
* Must be at least 18 years of age and not older than 55 years of age
* Must have been stable on a dose of Abilify, Risperdal, Seroquel, or Zyprexa for the past 8 weeks
* Women of childbearing potential must be using a medically accepted means of contraception
* Must be able to swallow capsules

Exclusion Criteria:

* Has serious health problems other than Schizophrenia
* Takes an antidepressant for depression
* Takes insulin for diabetes
* Have a history of alcohol or drug dependence (except for nicotine and caffeine) within the past 6 months

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult

CONTACTS AND LOCATIONS:
Locations (20):
- United States (20):
  - "For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at (1-877-285-4559) or speak with your personal physician.", Cerritos, California
  - "For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at (1-877-285-4559) or speak with your personal physician., Chula Vista, California
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY(1-877-285-4559) or speak with your personal physician., Garden Grove, California
  - "For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at (1-877-285-4559) or speak with your personal physician.", San Diego, California
  - "For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at (1-877-285-4559) or speak with your personal physician.", New Haven, Connecticut
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY(1-877-285-4559) or speak with your personal physician., New Haven, Connecticut
  - "For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at (1-877-285-4559) or speak with your personal physician.", Atlanta, Georgia
  - "For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at (1-877-285-4559) or speak with your personal physician.", Chicago, Illinois
  - "For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at (1-877-285-4559) or speak with your personal physician.", Indianapolis, Indiana
  - "For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at (1-877-285-4559) or speak with your personal physician.", Iowa City, Iowa
  - "For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at (1-877-285-4559) or speak with your personal physician.", Minneapolis, Minnesota
  - "For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at (1-877-285-4559) or speak with your personal physician.", Lebanon, New Hampshire
  - "For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at (1-877-285-4559) or speak with your personal physician.", New York, New York
  - "For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at (1-877-285-4559) or speak with your personal physician.", Butner, North Carolina
  - "For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at (1-877-285-4559) or speak with your personal physician.", Chapel Hill, North Carolina
  - "For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at (1-877-285-4559) or speak with your personal physician.", Okalahoma City, Oklahoma
  - "For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at (1-877-285-4559) or speak with your personal physician.", Austin, Texas
  - "For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at (1-877-285-4559) or speak with your personal physician.", Irving, Texas
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY(1-877-285-4559) or speak with your personal physician., Irving, Texas
  - "For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at (1-877-285-4559) or speak with your personal physician.", San Antonio, Texas